CLINICAL TRIAL: NCT02912468
Title: A Randomized, 24-Week Treatment, Double-blind, Placebo-controlled Efficacy and Safety Study of Dupilumab 300 mg Every Other Week, in Patients With Bilateral Nasal Polyposis on a Background Therapy With Intranasal Corticosteroids
Brief Title: A Controlled Clinical Study of Dupilumab in Patients With Bilateral Nasal Polyps
Acronym: SINUS-24
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC14146; 2015-003101-42 (EudraCT Number); U1111-1178-5390 (Other: UTN)
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Chronic Rhinosinusitis Phenotype With Nasal Polyps (CRSwNP)
Keywords: Nasal polyposis, Chronic rhinosinusitis, Intranasal corticosteroids, Dupilumab, Human monoclonal antibody
MeSH Terms: conditions — Nasal Polyps | interventions — dupilumab; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Dupilumab and placebo were provided in matching 2 milliliter (mL) pre-filled syringes. To protect the blind, each treatment kit was prepared such that the dupilumab dose and its corresponding placebo volume were identical and indistinguishable and were labelled with a treatment kit number.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for dupilumab), 1 subcutaneous (SC) injection every 2 weeks (q2w) from Day 1 of Week 0 up to Week 24 added to background therapy of intranasal mometasone furoate nasal spray (MFNS) at stable dose.
  Interventions: Drug: Placebo; Drug: Mometasone furoate 50 micrograms
- Dupilumab 300 mg (Experimental): Dupilumab 300 mg SC injection q2w from Day 1 of Week 0 up to Week 24 added to background therapy of intranasal MFNS at stable dose.
  Interventions: Drug: Dupilumab SAR231893 (REGN668); Drug: Mometasone furoate 50 micrograms

INTERVENTIONS:
Drug: Dupilumab SAR231893 (REGN668) — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: Dupilumab 300 mg
Drug: Placebo — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: Placebo
Drug: Mometasone furoate 50 micrograms — Pharmaceutical form: Suspension (Nasal spray)
  Route of administration: Intranasal
  Other Names: NASONEX®

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab 300 milligram (mg) every 2 weeks (q2w) compared to placebo on a background of mometasone furoate nasal spray (MFNS) in reducing nasal congestion/obstruction (NC) severity and endoscopic nasal polyp score (NPS) in participants with bilateral nasal polyposis (NP). In addition for Japan participants, reduction in computed tomography (CT) scan opacification of the sinuses was a coprimary objective.

Secondary Objectives:

* To evaluate the efficacy of dupilumab in improving total symptoms score (TSS).
* To evaluate the efficacy of dupilumab in improving sense of smell.
* To evaluate the efficacy of dupilumab in reducing CT scan opacification of the sinuses (primary objective for Japan).
* To evaluate ability of dupilumab in reducing proportion of participants requiring treatment with systemic corticosteroids or NP surgery.
* To evaluate the effect of dupilumab on participant reported outcomes and health related quality of life outcome by sinonasal outcome test-22 (SNOT-22).
* To evaluate the effect of dupilumab in the subgroups of participants with prior surgery and co-morbid asthma (including non-steroid antiinflammatory drug [NSAID] exacerbated respiratory disease [ERD]).
* To evaluate residual effect in follow up.
* To evaluate the safety of dupilumab in participants with bilateral NP.
* To evaluate functional dupilumab concentrations (systemic exposure) and incidence of treatment-emergent anti-drug antibodies.

DETAILED DESCRIPTION:
The total study duration per participant was expected to be up to 52 weeks that consisted of a 4-weeks run-in period, 24-weeks treatment period, and a 24-weeks post treatment period.

ELIGIBILITY:
Inclusion criteria:

* Participants with bilateral sinonasal polyposis that despite prior treatment with systemic corticosteroids (SCS) anytime within the past 2 years; and/or had a medical contraindication / intolerance to SCS; and/or had prior surgery for NP at the screening visit, had:
* An endoscopic bilateral NPS of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity).
* Ongoing symptoms (for at least 8 weeks prior to Visit [V] 1) of nasal congestion/blockage/obstruction with moderate or severe symptom severity (score 2 or 3) at V1 and a weekly average severity of greater than 1 at the time of randomization (V2), and another symptom such as loss of smell, rhinorrhea (anterior/posterior).
* Signed written informed consent.

Exclusion criteria:

* Participants <18 years of age.
* Participants who were previously treated in dupilumab studies.
* Participants who had taken:
* Biologic therapy/systemic immunosuppressant to treat inflammatory disease or autoimmune disease (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, etc.) within 2 months before V1 or 5 half-lives, whichever was longer.
* Any experimental monoclonal antibody (mAB) within 5 half-lives or within 6 months before V1 if the half-life was unknown.
* Anti-immunoglobulin E (IgE) therapy (omalizumab) within 130 days prior to V1.
* Participants who received leukotriene antagonists/modifiers at V1 unless they were on a continuous treatment for at least 30 days prior to V1.
* Initiated allergen immunotherapy within 3 months prior to V1 or planned to begin therapy or changed its dose during the run-in period or the randomized treatment period.
* Participants who undergone any intranasal and/or sinus surgery (including polypectomy) within 6 months prior to V1.
* Participants who had a sinonasal or sinus surgery changing the lateral wall structure of the nose making impossible the evaluation of NPS.
* Participants with conditions/concomitant diseases making them nonevaluable at V1 or for the primary efficacy endpoint such as:
* Antrochoanal polyps;
* Nasal septal deviation that would occlude at least one nostril;
* Acute sinusitis, nasal infection or upper respiratory infection;
* Ongoing rhinitis medicamentosa;
* Allergic granulomatous angiitis (Churg-Strauss syndrome), granulomatosis with polyangiitis (Wegener's granulomatosis), Young's syndrome, Kartagener's syndrome or other dyskinetic ciliary syndromes, concomitant cystic fibrosis;
* Radiologic suspicion, or confirmed invasive or expansive fungal rhinosinusitis.
* Participants with nasal cavity malignant tumor and benign tumors (eg, papilloma, blood boil, etc).
* Participants with forced expiratory volume in 1 second (FEV1) 50% or less (of predicted normal).
* Participants who received concomitant treatment prohibited in the study.
* Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit.
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Positive with hepatitis B surface antigen (HBsAg) or hepatitis C antibody at the screening visit.
* Active chronic or acute infection requiring systemic treatment within 2 weeks before the baseline visit.
* Known or suspected history of immunosuppression.
* Pregnant or breastfeeding women, or women planned to become pregnant or breastfeed during the study.
* Women unwilling to use adequate birth control, if of reproductive potential and sexually active.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (76):
- United States (18):
  - Investigational Site Number 8400009, Long Beach, California
  - Investigational Site Number 8400004, Orange, California
  - Investigational Site Number 8400014, San Diego, California
  - Investigational Site Number 8400002, Stockton, California
  - Investigational Site Number 8400016, Centennial, Colorado
  - Investigational Site Number 8400013, Tampa, Florida
  - Investigational Site Number 8400022, West Des Moines, Iowa
  - Investigational Site Number 8400007, Boston, Massachusetts
  - Investigational Site Number 8400005, Rochester, Minnesota
  - Investigational Site Number 8400021, St Louis, Missouri
  - Investigational Site Number 8400008, Winston-Salem, North Carolina
  - Investigational Site Number 8400019, Tulsa, Oklahoma
  - Investigational Site Number 8400020, Medford, Oregon
  - Investigational Site Number 8400018, Charleston, South Carolina
  - Investigational Site Number 8400003, Nashville, Tennessee
  - Investigational Site Number 8400001, Dallas, Texas
  - Investigational Site Number 8400015, Norfolk, Virginia
  - Investigational Site Number 8400010, Milwaukee, Wisconsin
- Bulgaria (3):
  - Investigational Site Number 1000003, Plovdiv
  - Investigational Site Number 1000002, Sofia
  - Investigational Site Number 1000001, Sofia
- Czechia (3):
  - Investigational Site Number 2030001, Hradec Králové
  - Investigational Site Number 2030002, Pardubice
  - Investigational Site Number 2030004, Prague
- France (7):
  - Investigational Site Number 2500005, La Roche-sur-Yon
  - Investigational Site Number 2500007, Lille
  - Investigational Site Number 2500003, Lyon
  - Investigational Site Number 2500001, Montpellier
  - Investigational Site Number 2500006, Nantes
  - Investigational Site Number 2500002, Toulouse
  - Investigational Site Number 2500004, Vandœuvre-lès-Nancy
- Germany (3):
  - Investigational Site Number 2760001, Berlin
  - Investigational Site Number 2760003, München
  - Investigational Site Number 2760002, Münster
- Hungary (7):
  - Investigational Site Number 3480006, Budapest
  - Investigational Site Number 3480007, Budapest
  - Investigational Site Number 3480004, Budapest
  - Investigational Site Number 3480003, Budapest
  - Investigational Site Number 3480005, Debrecen
  - Investigational Site Number 3480002, Pécs
  - Investigational Site Number 3480001, Szeged
- Italy (7):
  - Investigational Site Number 3800007, Bologna
  - Investigational Site Number 3800002, Catania
  - Investigational Site Number 3800004, Milan
  - Investigational Site Number 3800006, Milan
  - Investigational Site Number 3800001, Pisa
  - Investigational Site Number 3800005, Rozzano
  - Investigational Site Number 3800003, Varese
- Investigational Site Number 5280001, Amsterdam, Netherlands
- Poland (3):
  - Investigational Site Number 6160002, Katowice
  - Investigational Site Number 6160001, Lodz
  - Investigational Site Number 6160003, Warsaw
- Romania (6):
  - Investigational Site Number 6420007, Brasov
  - Investigational Site Number 6420013, Brasov
  - Investigational Site Number 6420003, Bucharest
  - Investigational Site Number 6420009, Cluj-Napoca
  - Investigational Site Number 6420008, Craiova
  - Investigational Site Number 6420010, Târgu Mureş
- Russia (6):
  - Investigational Site Number 6430004, Moscow
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430002, Saint Petersburg
  - Investigational Site Number 6430001, Saint Petersburg
  - Investigational Site Number 6430007, Saint Petersburg
  - Investigational Site Number 6430006, Yaroslavl
- Ukraine (6):
  - Investigational Site Number 8040002, Ivano-Frankivsk
  - Investigational Site Number 8040004, Kharkiv
  - Investigational Site Number 8040005, Kyiv
  - Investigational Site Number 8040006, Kyiv
  - Investigational Site Number 8040001, Poltava
  - Investigational Site Number 8040008, Ternopil
- United Kingdom (6):
  - Investigational Site Number 8260001, Bradford
  - Investigational Site Number 8260002, Dundee
  - Investigational Site Number 8260007, Great Yarmouth
  - Investigational Site Number 8260006, London
  - Investigational Site Number 8260004, Stockport
  - Investigational Site Number 8260005, Wigan

IPD SHARING:
Plan to Share IPD: No
Not yet available

REFERENCES:
- [Derived] Lane AP, Mullol J, Hopkins C, Fokkens WJ, Lee SE, Msihid J, Nash S, Sacks H, Borsos K, Kamat S, Rowe PJ, Deniz Y, Jacob-Nara JA. Dupilumab improves sense of smell and clinical outcomes in patients with severe chronic rhinosinusitis with nasal polyps with anosmia. Curr Med Res Opin. 2025 Jan;41(1):53-59. doi: 10.1080/03007995.2024.2434083. Epub 2024 Dec 14. PMID 39618256
- [Derived] Bachert C, Khan AH, Hopkins C, Han JK, Fokkens WJ, Mannent LP, Msihid J, Borsos K, Kamat S, Nash S, Sacks H, Rowe PJ, Deniz Y, Jacob-Nara JA. Mild and symptom-free months in patients with chronic rhinosinusitis with nasal polyps treated with dupilumab. Ann Allergy Asthma Immunol. 2025 Jan;134(1):61-69.e12. doi: 10.1016/j.anai.2024.09.015. Epub 2024 Sep 28. PMID 39343385
- [Derived] Hopkins C, Mullol J, Khan AH, Lee SE, Wagenmann M, Hellings P, Fokkens W, Msihid J, Nair R, Kamat S, Nash S, Radwan A, Jacob-Nara JA, Deniz Y, Rowe PJ. Impact of Dupilumab on Sinonasal Symptoms and Outcomes in Severe Chronic Rhinosinusitis With Nasal Polyps. Otolaryngol Head Neck Surg. 2024 Apr;170(4):1173-1182. doi: 10.1002/ohn.627. Epub 2023 Dec 29. PMID 38156522
- [Derived] Maspero JF, Bachert C, Martinez FJ, Hanania NA, Ortiz B, Patel N, Mannent LP, Praestgaard A, Pandit-Abid N, Siddiqui S, Hardin M. Clinical Efficacy among Patients with Chronic Rhinosinusitis with Nasal Polyps and Clinical Features of Obstructive Lung Disease: Post Hoc Analysis of the Phase III SINUS-24 and SINUS-52 Studies. J Asthma Allergy. 2023 Mar 31;16:333-342. doi: 10.2147/JAA.S357393. eCollection 2023. PMID 37026112
- [Derived] Peters AT, Soler ZM, Kern RC, Heffler E, Maspero JF, Crampette L, Fujieda S, Lane AP, Zhang H, Nash S, Khan AH, Siddiqui S, Jacob-Nara JA, Rowe P, Deniz Y. Improvement in patient-reported "taste" and association with smell in dupilumab-treated patients with severe chronic rhinosinusitis with nasal polyps from the SINUS-24 and SINUS-52 trials. Clin Exp Allergy. 2022 Sep;52(9):1105-1109. doi: 10.1111/cea.14194. Epub 2022 Jul 12. No abstract available. PMID 35775319
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Bachert C, Peters AT, Heffler E, Han JK, Olze H, Pfaar O, Chuang CC, Rout R, Attre R, Goga L, Jacob-Nara JA, Rowe PJ, Deniz Y, Chen Z, Kamat S, Siddiqui S. Responder analysis to demonstrate the effect of targeting type 2 inflammatory mechanisms with dupilumab across objective and patient-reported endpoints for patients with severe chronic rhinosinusitis with nasal polyps in the SINUS-24 and SINUS-52 studies. Clin Exp Allergy. 2022 Feb;52(2):244-249. doi: 10.1111/cea.14051. No abstract available. PMID 35092110
- [Derived] Lee SE, Hopkins C, Mullol J, Msihid J, Guillemin I, Amin N, Mannent LP, Li Y, Siddiqui S, Chuang CC, Kamat S, Khan AH. Dupilumab improves health related quality of life: Results from the phase 3 SINUS studies. Allergy. 2022 Jul;77(7):2211-2221. doi: 10.1111/all.15222. Epub 2022 Feb 1. PMID 35034364
- [Derived] Bachert C, Corren J, Lee SE, Zhang H, Harel S, Cunoosamy D, Khan AH, Jacob-Nara JA, Siddiqui S, Nash S, Rowe PJ, Deniz Y. Dupilumab efficacy and biomarkers in chronic rhinosinusitis with nasal polyps: Association between dupilumab treatment effect on nasal polyp score and biomarkers of type 2 inflammation in patients with chronic rhinosinusitis with nasal polyps in the phase 3 SINUS-24 and SINUS-52 trials. Int Forum Allergy Rhinol. 2022 Sep;12(9):1191-1195. doi: 10.1002/alr.22964. Epub 2022 Jan 31. No abstract available. PMID 34970860
- [Derived] Hellings PW, Peters AT, Chaker AM, Heffler E, Zhang H, Praestgaard A, Nash S, Khan AH, Siddiqui S, Jacob-Nara JA, Rowe PJ, Deniz Y. Rapid and sustained effects of dupilumab in severe chronic rhinosinusitis with nasal polyps. Int Forum Allergy Rhinol. 2022 Jul;12(7):958-962. doi: 10.1002/alr.22944. Epub 2022 Jan 23. No abstract available. PMID 34911163
- [Derived] Han JK, Bachert C, Lee SE, Hopkins C, Heffler E, Hellings PW, Peters AT, Kamat S, Whalley D, Qin S, Nelson L, Siddiqui S, Khan AH, Li Y, Mannent LP, Guillemin I, Chuang CC. Estimating Clinically Meaningful Change of Efficacy Outcomes in Inadequately Controlled Chronic Rhinosinusitis with Nasal Polyposis. Laryngoscope. 2022 Feb;132(2):265-271. doi: 10.1002/lary.29888. Epub 2021 Dec 1. PMID 34850966
- [Derived] Chuang CC, Guillemin I, Bachert C, Lee SE, Hellings PW, Fokkens WJ, Duverger N, Fan C, Daizadeh N, Amin N, Mannent LP, Khan AH, Kamat S. Dupilumab in CRSwNP: Responder Analysis Using Clinically Meaningful Efficacy Outcome Thresholds. Laryngoscope. 2022 Feb;132(2):259-264. doi: 10.1002/lary.29911. Epub 2021 Nov 24. PMID 34817082
- [Derived] Mullol J, Laidlaw TM, Bachert C, Mannent LP, Canonica GW, Han JK, Maspero JF, Picado C, Daizadeh N, Ortiz B, Li Y, Ruddy M, Laws E, Amin N. Efficacy and safety of dupilumab in patients with uncontrolled severe chronic rhinosinusitis with nasal polyps and a clinical diagnosis of NSAID-ERD: Results from two randomized placebo-controlled phase 3 trials. Allergy. 2022 Apr;77(4):1231-1244. doi: 10.1111/all.15067. Epub 2021 Oct 1. PMID 34459002
- [Derived] Khan AH, Reaney M, Guillemin I, Nelson L, Qin S, Kamat S, Mannent L, Amin N, Whalley D, Hopkins C. Development of Sinonasal Outcome Test (SNOT-22) Domains in Chronic Rhinosinusitis With Nasal Polyps. Laryngoscope. 2022 May;132(5):933-941. doi: 10.1002/lary.29766. Epub 2021 Aug 26. PMID 34437720
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614
- [Derived] Hopkins C, Wagenmann M, Bachert C, Desrosiers M, Han JK, Hellings PW, Lee SE, Msihid J, Radwan A, Rowe P, Amin N, Deniz Y, Ortiz B, Mannent LP, Rout R. Efficacy of dupilumab in patients with a history of prior sinus surgery for chronic rhinosinusitis with nasal polyps. Int Forum Allergy Rhinol. 2021 Jul;11(7):1087-1101. doi: 10.1002/alr.22780. Epub 2021 Feb 21. PMID 33611847
- [Derived] Peters AT, Han JK, Hellings P, Heffler E, Gevaert P, Bachert C, Xu Y, Chuang CC, Neupane B, Msihid J, Mannent LP, Guyot P, Kamat S. Indirect Treatment Comparison of Biologics in Chronic Rhinosinusitis with Nasal Polyps. J Allergy Clin Immunol Pract. 2021 Jun;9(6):2461-2471.e5. doi: 10.1016/j.jaip.2021.01.031. Epub 2021 Feb 4. PMID 33548517
- [Derived] Laidlaw TM, Bachert C, Amin N, Desrosiers M, Hellings PW, Mullol J, Maspero JF, Gevaert P, Zhang M, Mao X, Khan AH, Kamat S, Patel N, Graham NMH, Ruddy M, Staudinger H, Mannent LP. Dupilumab improves upper and lower airway disease control in chronic rhinosinusitis with nasal polyps and asthma. Ann Allergy Asthma Immunol. 2021 May;126(5):584-592.e1. doi: 10.1016/j.anai.2021.01.012. Epub 2021 Jan 16. PMID 33465455
- [Derived] Bachert C, Han JK, Desrosiers M, Hellings PW, Amin N, Lee SE, Mullol J, Greos LS, Bosso JV, Laidlaw TM, Cervin AU, Maspero JF, Hopkins C, Olze H, Canonica GW, Paggiaro P, Cho SH, Fokkens WJ, Fujieda S, Zhang M, Lu X, Fan C, Draikiwicz S, Kamat SA, Khan A, Pirozzi G, Patel N, Graham NMH, Ruddy M, Staudinger H, Weinreich D, Stahl N, Yancopoulos GD, Mannent LP. Efficacy and safety of dupilumab in patients with severe chronic rhinosinusitis with nasal polyps (LIBERTY NP SINUS-24 and LIBERTY NP SINUS-52): results from two multicentre, randomised, double-blind, placebo-controlled, parallel-group phase 3 trials. Lancet. 2019 Nov 2;394(10209):1638-1650. doi: 10.1016/S0140-6736(19)31881-1. Epub 2019 Sep 19. PMID 31543428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were involved in the study from 05 December 2016 to 05 July 2018 at 67 active centers in 13 countries. A total of 506 participants were screened, of which 276 participants were enrolled and randomized to receive dupilumab 300 mg or placebo. A total of 230 participants failed screening mainly due to failure to meet inclusion criteria.
Pre-assignment Details: Randomization was stratified by the presence of comorbid asthma and/or non-steroidal anti-inflammatory drug exacerbated respiratory disease (NSAID-ERD), prior nasal polyposis (NP) surgery (yes or no), and country.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg
Started | 133 | 143
Treated | 133 | 142
Safety Population (1 participant of placebo arm received 1 dose of dupilumab: counted in dupilumab for safety analysis.) | 132 | 143
Completed | 124 | 138
Not Completed | 9 | 5
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Randomized and not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized participants, which included any participant who was allocated to a randomized treatment regardless of whether any treatment kit was used.
Groups:
- Placebo: Placebo (for dupilumab), 1 SC injection q2w from Day 1 of Week 0 up to Week 24 added to background therapy of intranasal MFNS at stable dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg | Total
Number analyzed (Participants) | 133 | 143 | 276
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.83 (13.21) | 50.17 (13.59) | 50.49 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 55 | 118
  Male | 70 | 88 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: "Number analyzed" = Number of participants evaluable for the specified baseline measure.
  Participants
    number analyzed (Participants) | 131 | 143 | 274
    Hispanic or Latino | 1 | 5 | 6
    Not Hispanic or Latino | 130 | 138 | 268
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 126 | 138 | 264
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Nasal Congestion/Obstruction (NC) Symptom Severity Score [Mean (Standard Deviation); unit: score on a scale] — NC symptom severity was assessed by the participants on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity.
  score on a scale | 2.45 (0.55) | 2.26 (0.57) | 2.35 (0.57)
Nasal Polyp Score (NPS) [Mean (Standard Deviation); unit: score on a scale] — NPS was the sum of right and left nostril scores, as evaluated by means of nasal endoscopy. For each nostril, NPS was graded based on polyp size from 0 to 4 (0 = no polyps to 4 = large polyps causing complete obstruction of the inferior nasal cavity), with a lower score indicating smaller-sized polyps. Total NPS was the sum of right and left nostril scores and ranges from 0 (no polyps) to 8 (large polyps), with higher score representing more severe disease. Population: "Number analyzed" = Number of participants evaluable for the specified baseline measure.
  score on a scale
    number analyzed (Participants) | 132 | 143 | 275
    (all) | 5.86 (1.31) | 5.64 (1.23) | 5.75 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 24 in Nasal Congestion/Obstruction Symptom Severity Score
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Least squares (LS) means and standard error (SE) were obtained from Analysis of covariance (ANCOVA) model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 24
Population: The analysis was performed on intent-to-treat (ITT) population which included all randomized participants who were analyzed according to the treatment group allocated by randomization.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale | -0.45 (0.07) | -1.34 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg; Data were analyzed using a hybrid method of the worst-observation carried forward (WOCF) and multiple imputation (MI). The imputed completed data were analyzed by fitting ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. Statistical inference obtained from all imputed data was combined using Rubin's rule; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -0.89, 95% CI 2-sided [-1.07 to -0.71]

2. Primary Outcome: Change From Baseline at Week 24 in Nasal Polyp Score
Description: NPS: sum of right, left nostril scores, evaluated by nasal endoscopy. For each nostril, NPS was graded based on polyp size from 0 = no polyps to 4 = large polyps causing complete obstruction of inferior nasal cavity; lower score = smaller-sized polyps. Total NPS: sum of right and left nostril scores; ranges from 0 (no polyps) to 8 (large polyps), higher score = more severe disease. NPS was assessed by centralized, blinded, independent review of the nasal endoscopy video recordings. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 24
Population: The analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 132 | 143
score on a scale | 0.17 (0.15) | -1.89 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg; Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates. Statistical inference obtained from all imputed data was combined using Rubin's rule; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -2.06, 95% CI 2-sided [-2.43 to -1.69]

3. Secondary Outcome: Change From Baseline at Week 24 in Opacification of Sinuses Measured by Lund-Mackay (LMK) Score
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview. NOTE: For Japan regulatory submission only, this endpoint is not included as a secondary outcome measure and is instead one of the co-primary outcome measures.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 129 | 141
score on a scale | -0.74 (0.37) | -8.18 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Hierarchical testing procedure was used to control type I error. For regions outside of Japan, this first secondary endpoint was not tested unless both co-primary endpoints were significant at the 0.05 level. Hierarchical testing continued only when previous endpoint was statistically significant. For Japan submission, LMK was instead a co-primary endpoint which also had to be met before secondary endpoints were tested in the hierarchy. Last endpoint in hierarchy is Week 24 SNOT-22; p < .0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -7.44, 95% CI 2-sided [-8.35 to -6.53]

4. Secondary Outcome: Change From Baseline at Week 24 in Total Symptom Score (TSS)
Description: The TSS was the sum of participant-assessed nasal symptom scores for nasal congestion/obstruction, decreased/loss of sense of smell, and rhinorrhea (anterior/posterior nasal discharge), each accessed on 0-3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms). Total score ranged from 0 (no symptoms) to 9 (severe symptoms). Higher score indicated more severe symptoms. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 24
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale | -1.17 (0.17) | -3.77 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Testing according to the hierarchical testing procedure (only performed if previous outcome measures were statistically significant); p < .0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -2.61, 95% CI 2-sided [-3.04 to -2.17]

5. Secondary Outcome: Change From Baseline at Week 24 in the University of Pennsylvania Smell Identification Test (UPSIT) Score
Description: The UPSIT was a 40-item test to measure the individual's ability to detect odors. Total score ranges from 0 (anosmia) to 40 (normal sense of smell), lower score indicated severe smell loss. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 24
Population: The analysis was performed on ITT. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 140
score on a scale | 0.70 (0.71) | 11.26 (0.67)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < .0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = 10.56, 95% CI 2-sided [8.79 to 12.34]

6. Secondary Outcome: Change From Baseline at Week 24 in Severity of Decreased/Loss of Smell as Assessed by Participant Daily
Description: The severity of decreased/loss of sense of smell was reported by the participants using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), higher score indicated more severe symptoms. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 24
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale | -0.29 (0.07) | -1.41 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < .0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -1.12, 95% CI 2-sided [-1.31 to -0.93]

7. Secondary Outcome: Change From Baseline at Week 24 in 22-item Sino-nasal Outcome Test (SNOT-22) Scores
Description: The SNOT-22 is a validated questionnaire that was used to assess the impact of chronic rhinosinusitis phenotype with nasal polyps (CRSwNP) on health-related quality of life (HRQoL). It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life. LS means and SE were obtained from ANCOVA model described in Statistical Analysis Overview.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 131 | 137
score on a scale | -9.31 (1.62) | -30.43 (1.54)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < .0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -21.12, 95% CI 2-sided [-25.17 to -17.06]

8. Secondary Outcome: Rescue Treatment Use: Estimate of Percentage of Participants With >=1 Event by Week 24 Obtained Using Kaplan-Meier Method
Description: Rescue treatment was defined as usage of systemic corticosteroids (SCS) or NP surgery (actual or planned) during the treatment period. Rescue treatment included:
  * SCS: Betamethasone, dexamethasone, dexamethasone sodium phosphate, Hydrocortisone sodium succinate, methylprednisolone, prednisolone, prednisolone metasulfobenzoate sodium, prednisone, and triamcinolone.
  * Sino-nasal surgery for nasal polyps when there was worsening of signs and/or symptoms during the study.
  Estimate of percentage of participants with event by Week 24 was obtained using Kaplan-Meier method.
Time Frame: Baseline up to Week 24
Population: The analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants with event
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
percentage of participants with event
  SCS treatment | 18.9 [12.7 to 26.0] | 6.5 [3.2 to 11.5]
  NP surgery | 7.5 [3.7 to 13.2] | 2.1 [0.6 to 5.6]

9. Secondary Outcome: Change From Baseline at Week 24 in Visual Analogue Scale (VAS) for Rhinosinusitis
Description: The VAS for rhinosinusitis was used to evaluate the total disease severity. The participants were asked to indicate on a 10 centimeters (cm) VAS the answer to the question, "How troublesome are your symptoms of your rhinosinusitis?" The range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome), where higher score indicated worse thinkable troublesome. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 130 | 136
centimeters | -1.34 (0.24) | -4.54 (0.23)

10. Secondary Outcome: Change From Baseline at Week 24 in Nasal Peak Inspiratory Flow (NPIF)
Description: NPIF evaluation represented a physiologic measure of the air flow through both nasal cavities during forced inspiration expressed in liters per minute. Higher NPIF values are indicative of better nasal air flow. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 24
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: liters per minute
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
liters per minute | 14.09 (3.97) | 54.50 (3.73)

11. Secondary Outcome: Change From Baseline at Week 24 in Rhinorrhea Daily Symptom Score
Description: Rhinorrhea was reported by the participants using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), where higher scores indicated more severe symptoms. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 24
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale | -0.42 (0.06) | -1.04 (0.06)

12. Secondary Outcome: Change From Baseline at Week 24 in Forced Expiratory Volume in 1 Second (FEV1) for Participants With Asthma
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants which included all randomized participants with asthma.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 79 | 82
liters | -0.06 (0.05) | 0.15 (0.05)

13. Secondary Outcome: Change From Baseline at Week 24 in Asthma Control Questionnaire-6 (ACQ-6) Scores for Participants With Asthma
Description: ACQ-6 had 6 questions which assessed the most common asthma symptoms (woken by asthma, symptoms on waking, activity limitation, shortness of breath, wheezing, puffs/inhalations use). Participants were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale ranged from 0 = no impairment to 6 = maximum impairment. The ACQ-6 score was the mean of the scores of all 6 questions and therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled), with higher scores indicated lower asthma control. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with the corresponding baseline value, treatment group, prior surgery, and regions as covariates.
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants which included all randomized participants with asthma and had available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 76 | 75
score on a scale | -0.24 (0.10) | -1.00 (0.10)

14. Secondary Outcome: Change From Baseline at Weeks 28, 32, 36, 40, 44 and 48 in Nasal Congestion Symptom Severity Score (Assessments Performed 4-24 Weeks After End of Treatment)
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48 (Post-baseline assessments performed 4-24 weeks after end of treatment)
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale
  Week 28 | -0.48 (0.07) | -1.36 (0.07)
  Week 32 | -0.50 (0.07) | -1.33 (0.07)
  Week 36 | -0.53 (0.07) | -1.05 (0.07)
  Week 40 | -0.51 (0.08) | -0.83 (0.07)
  Week 44 | -0.49 (0.08) | -0.77 (0.07)
  Week 48 | -0.52 (0.08) | -0.77 (0.07)

15. Secondary Outcome: Change From Baseline at Weeks 36 and 48 in Nasal Polyp Score (Assessments Performed 12 and 24 Weeks After End of Treatment)
Description: NPS was the sum of right and left nostril scores, as evaluated by means of nasal endoscopy. For each nostril, NPS was graded based on polyp size from 0 to 4 (0 = no polyps to 4 = large polyps causing complete obstruction of the inferior nasal cavity), with a lower score indicating smaller-sized polyps. Total NPS was the sum of right and left nostril scores and ranges from 0 (no polyp) to 8 (large polyp), with highest score representing more severe disease. NPS was assessed by centralized, blinded, independent review of the nasal endoscopy video recordings. Data were analyzed using a hybrid method of the WOCF and MI. LS mean and SE were obtained from ANCOVA model.
Time Frame: Baseline, Week 36, Week 48 (post-baseline assessments performed 12 and 24 weeks after end of treatment)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 132 | 143
score on a scale
  Week 36 | -0.06 (0.14) | -0.99 (0.13)
  Week 48 | 0.14 (0.13) | -0.66 (0.12)

16. Secondary Outcome: Change From Baseline at Week 48 in Opacification of Sinuses Measured by Lund-Mackay Score (Assessment Performed 24 Weeks After End of Treatment)
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 48 (Post-baseline assessment performed 24 weeks after end of treatment)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 129 | 141
score on a scale | -0.82 (0.38) | -2.62 (0.36)

17. Secondary Outcome: Change From Baseline at Weeks 28, 32, 36, 40, 44 and 48 in Total Symptom Score (Assessments Performed 4-24 Weeks After End of Treatment)
Description: The TSS was the sum of participant-assessed nasal symptom scores for NC/obstruction, decreased/loss of sense of smell, and rhinorrhea (anterior/posterior nasal discharge), each accessed on 0-3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms). Total score ranged from 0 (no symptoms) to 9 (severe symptoms). Higher score indicated more severe symptoms. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: as for outcome 14
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale
  Week 28 | -1.18 (0.17) | -3.84 (0.16)
  Week 32 | -1.25 (0.17) | -3.64 (0.17)
  Week 36 | -1.31 (0.18) | -2.91 (0.17)
  Week 40 | -1.27 (0.18) | -2.28 (0.17)
  Week 44 | -1.20 (0.18) | -2.09 (0.17)
  Week 48 | -1.28 (0.19) | -2.05 (0.18)

18. Secondary Outcome: Change From Baseline at Week 48 in University of Pennsylvania Smell Identification Test (Assessment Performed 24 Weeks After End of Treatment)
Description: The UPSIT was a 40-item test to measure the individual's ability to detect odors. Total score ranges from 0 (anosmia) to 40 (normal sense of smell), lower score indicated severe smell loss. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 48 (Post-baseline assessment performed 24 weeks after end of treatment)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 140
score on a scale | 0.21 (0.77) | 4.20 (0.73)

19. Secondary Outcome: Change From Baseline at Weeks 28, 32, 36, 40, 44 and 48 in Severity of Decreased/Loss of Smell as Assessed by Participant Daily (Assessments Performed 4-24 Weeks After End of Treatment)
Description: The severity of decreased/loss of sense of smell was reported by the participants using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), higher score indicated more severe symptoms. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: as for outcome 14
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale
  Week 28 | -0.28 (0.08) | -1.45 (0.07)
  Week 32 | -0.31 (0.08) | -1.36 (0.07)
  Week 36 | -0.33 (0.08) | -1.07 (0.07)
  Week 40 | -0.30 (0.07) | -0.83 (0.07)
  Week 44 | -0.28 (0.07) | -0.74 (0.07)
  Week 48 | -0.30 (0.07) | -0.71 (0.06)

20. Secondary Outcome: Change From Baseline at Weeks 36 and 48 in 22-item Sino-nasal Outcome Test Scores (Assessments Performed 12 and 24 Weeks After End of Treatment)
Description: The SNOT-22 is a validated questionnaire that was used to assess the impact of CRSwNP on HRQoL. It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 36 and Week 48 (Post-baseline assessments performed 12 and 24 weeks after end of treatment)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 131 | 137
score on a scale
  Week 36 | -8.31 (1.75) | -20.87 (1.67)
  Week 48 | -8.36 (1.88) | -17.66 (1.80)

21. Secondary Outcome: Rescue Treatment Use: Estimate of Percentage of Participants With >=1 Event by Week 48 Obtained Using Kaplan-Meier Method
Description: Rescue treatment was defined as usage of SCS or NP surgery (actual or planned) during the study. Rescue treatment included:
  * SCS: Betamethasone, dexamethasone, dexamethasone sodium phosphate, Hydrocortisone sodium succinate, methylprednisolone, prednisolone, prednisolone metasulfobenzoate sodium, prednisone, and triamcinolone.
  * Sino-nasal surgery for nasal polyps when there was worsening of signs and/or symptoms during the study.
  Estimate of percentage of participants with event by Week 48 was obtained using Kaplan-Meier method.
Time Frame: Baseline up to Week 48
Population: The analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants with event
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
percentage of participants with event
  SCS treatment | 28.8 [21.4 to 36.7] | 21.4 [15.0 to 28.5]
  NP surgery | 12.5 [7.5 to 18.9] | 6.3 [2.9 to 11.4]

22. Secondary Outcome: Change From Baseline at Weeks 36 and 48 in Visual Analog Scale for Rhinosinusitis (Assessments Performed 12 and 24 Weeks After End of Treatment)
Description: The VAS for rhinosinusitis was used to evaluate the total disease severity. The participants were asked to indicate on a 10 cm VAS the answer to the question, "How troublesome are your symptoms of your rhinosinusitis?" The range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome), where higher score indicated worse thinkable troublesome. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 36 and Week 48 (Post-baseline assessments performed 12 and 24 weeks after end of treatment)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 130 | 136
centimeters
  Week 36 | -1.36 (0.26) | -3.02 (0.25)
  Week 48 | -1.17 (0.25) | -2.42 (0.24)

23. Secondary Outcome: Change From Baseline at Weeks 28, 32, 36, 40, 44 and 48 in Rhinorrhea Daily Symptom Score (Assessments Performed 4-24 Weeks After End of Treatment)
Description: as for outcome 11
Time Frame: as for outcome 14
Population: The analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 133 | 143
score on a scale
  Week 28 | -0.42 (0.06) | -1.04 (0.06)
  Week 32 | -0.43 (0.06) | -0.97 (0.06)
  Week 36 | -0.44 (0.07) | -0.80 (0.06)
  Week 40 | -0.44 (0.07) | -0.63 (0.06)
  Week 44 | -0.41 (0.07) | -0.58 (0.06)
  Week 48 | -0.45 (0.07) | -0.58 (0.07)

24. Secondary Outcome: Change From Baseline at Week 48 in Forced Expiratory Volume in 1 Second for Participants With Asthma (Assessment Performed 24 Weeks After End of Treatment)
Description: as for outcome 12
Time Frame: Baseline, Week 48 (Post-baseline assessment performed 24 weeks after end of treatment)
Population: Analysis was performed on a subset of participants which included all randomized participants with asthma.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 79 | 82
liters | -0.11 (0.05) | -0.05 (0.05)

25. Secondary Outcome: Change From Baseline at Week 48 in Asthma Control Questionnaire-6 Scores for Participants With Asthma (Assessment Performed 24 Weeks After End of Treatment)
Description: as for outcome 13
Time Frame: Baseline, Week 48 (Post-baseline assessment performed 24 weeks after end of treatment)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 76 | 75
score on a scale | -0.09 (0.11) | -0.55 (0.11)

26. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and TEAEs Leading to Treatment Discontinuation
Description: An Adverse Event (AE) was defined as any untoward medical occurrence that did not necessarily have to have a causal relationship with the study treatment. TEAEs were defined as AEs that developed or worsened in grade or became serious during TEAE period which was defined as the period from the time of first dose of study drug until 98 days following the last administration of study drug. Serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.
Time Frame: Baseline up to 98 days following the last administration of study drug (up to 36 weeks)
Population: The analysis was performed on safety population which included all participants who received at least 1 dose or part of a dose of the Investigational Medicinal Product (IMP), analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 132 | 143
Participants
  Any TEAE | 93 | 93
  Any treatment emergent SAE | 19 | 6
  TEAE leading to treatment discontinuation | 3 | 5

27. Secondary Outcome: Functional Dupilumab Concentration in Serum
Time Frame: Baseline, Week 4, 8, 16, 24, 36, End of study (Week 48)
Population: Analysis performed on pharmacokinetic population, which included participants who received atleast 1 dose of IMP with atleast 1 evaluable functional IMP concentration. Here, 'number analyzed'=number of participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for placebo
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 142
nanogram/milliliter
  Baseline: number analyzed (Participants) | 139
  Baseline | 0.00 (0.00)
  Week 4: number analyzed (Participants) | 138
  Week 4 | 31267.18 (13008.16)
  Week 8: number analyzed (Participants) | 141
  Week 8 | 48306.73 (20621.18)
  Week 16: number analyzed (Participants) | 138
  Week 16 | 63958.12 (29822.30)
  Week 24: number analyzed (Participants) | 136
  Week 24 | 69224.11 (36933.70)
  Week 36: number analyzed (Participants) | 136
  Week 36 | 356.53 (1501.69)
  Week 48: number analyzed (Participants) | 138
  Week 48 | 39.00 (0.00)

28. Secondary Outcome: Number of Participants With Treatment-Emergent And Treatment-Boosted Anti-drug Antibodies (ADA) Response
Description: ADA response were categorized as: treatment emergent and treatment boosted response. 1) Treatment emergent was defined as a positive response in the ADA assay post first dose, when baseline results are negative or missing. 2) Treatment boosted was defined as: An ADA positive response in the assay post first dose that is greater-than or equal to 4-fold over baseline titer levels, when baseline results are positive.
Time Frame: Baseline to End of study (Week 48)
Population: The analysis was performed on ADA population which included participants who received at least 1 dose of IMP with at least one non-missing ADA assay result following the first dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 132 | 143
Participants
  With treatment-emergent ADA | 7 | 22
  With treatment-boosted ADA | 0 | 0

29. Secondary Outcome: Mean Total Systemic Corticosteroids Rescue Dose Prescribed During Treatment Period
Description: SCS included: Betamethasone, dexamethasone, dexamethasone sodium phosphate, hydrocortisone sodium succinate, methylprednisolone, prednisolone, prednisolone metasulfobenzoate sodium, prednisone, and triamcinolone. For every participant, total dose was calculated as (prescribed total daily dose*duration of SCS use). Then, mean of the total dose of 25 participants (placebo group) and 9 participants (Dupilumab group) was derived.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 25 | 9
milligrams | 366.07 (247.07) | 686.65 (1575.86)

30. Secondary Outcome: Total Systemic Corticosteroids Rescue Intake Duration: Average Duration Per Participant
Description: Rescue treatment was defined as usage of SCS or NP surgery (actual or planned) during the treatment period. SCS rescue intake duration was defined as the duration (in days) from start of SCS rescue medication till the end of SCS rescue treatment.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 25 | 9
days | 11.04 (6.79) | 23.33 (50.13)

31. Secondary Outcome: Change From Baseline at Week 24 in European Quality of Life 5 Dimension (EQ-5D) Visual Analog Scale Score
Description: The EQ-5D was a standardized HRQoL questionnaire consisting of EQ-5D descriptive system and EQ VAS. EQ-5D descriptive system comprised of 5 dimensions: mobility, selfcare, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. EQ-VAS recorded the participant's self-rated health on a vertical VAS that allowed them to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable).
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 130 | 136
score on a scale | 1.74 (1.54) | 12.00 (1.48)

32. Secondary Outcome: Change From Baseline at Week 24 in Nasal Congestion Symptom Severity Score: Subgroup of Participants With Asthma
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting ANCOVA model with corresponding baseline, treatment group, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants, which included all randomized participants with asthma.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 79 | 82
score on a scale | -0.36 (0.09) | -1.48 (0.09)

33. Secondary Outcome: Change From Baseline at Week 24 in Nasal Congestion Symptom Severity Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: NC symptom severity was assessed by the participants on a daily basis from Visit 1 and throughout the study using an e-diary on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms, with higher scores indicated more severity. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, and regions as covariates.
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants, which included all randomized participants with prior NP surgery history.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 99 | 99
score on a scale | -0.52 (0.09) | -1.41 (0.08)

34. Secondary Outcome: Change From Baseline at Week 24 in Nasal Polyp Score: Subgroup of Participants With Asthma
Description: NPS was the sum of right and left nostril scores, as evaluated by means of nasal endoscopy. For each nostril, NPS was graded from 0 to 4 (0 = no polyps to 4 = large polyps causing complete obstruction of the inferior nasal cavity), with a lower score indicating smaller-sized polyps. Total NPS was the sum of right and left nostril scores and ranges from 0 (no polyp) to 8 (large polyp), with highest score representing more severe disease. NPS was assessed by centralized, blinded, independent review of the nasal endoscopy video recordings. Data were analyzed using a hybrid method of the WOCF and MI. LS mean and SE were obtained from ANCOVA model.
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants, which included all randomized participants with asthma and had available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 78 | 82
score on a scale | 0.27 (0.20) | -1.89 (0.20)

35. Secondary Outcome: Change From Baseline at Week 24 in Nasal Polyp Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: as for outcome 34
Time Frame: Baseline, Week 24
Population: Analysis was performed on a subset of participants, which included all randomized participants with prior NP surgery history and had available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 98 | 99
score on a scale | 0.14 (0.18) | -1.86 (0.18)

36. Secondary Outcome: Change From Baseline at Week 24 in Opacification of Sinuses Measured by Lund Mackay Score: Subgroup of Participants With Asthma
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, prior surgery history, and regions as covariates.
Time Frame: Baseline, Week 24
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 78 | 81
score on a scale | -0.15 (0.47) | -7.97 (0.47)

37. Secondary Outcome: Change From Baseline at Week 24 in Opacification of Sinuses Measured by Lund Mackay Score: Subgroup of Participants With Prior Nasal Polyp Surgery
Description: The LMK scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses using following grading: 0 = normal, 1 = partial opacification, 2 = total opacification. The total score was the sum of scores from each side and ranges from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. Data were analyzed using a hybrid method of the WOCF and MI. The imputed completed data were analyzed by fitting an ANCOVA model with corresponding baseline, treatment group, asthma/NSAID-ERD status, and regions as covariates.
Time Frame: Baseline, Week 24
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 97 | 98
score on a scale | -0.39 (0.42) | -7.60 (0.41)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to end of study regardless of seriousness or relationship to investigational product. Time frame for reporting of TEAE was up to 36 weeks.
Description: Reported AEs are treatment emergent AEs that developed/worsened during the 'on treatment period' (from the first IMP administration to the last study drug administration + 98 days). Analysis was performed on safety population.
Arm/Group | Placebo | Dupilumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/143
Serious Adverse Events (participants affected / at risk) | 19/132 | 6/143
Other Adverse Events (participants affected / at risk) | 61/132 | 55/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | Dupilumab 300 mg (N=143)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eosinophilic Granulomatosis With Polyangiitis (Immune system disorders) | 1 (1) | 1 (1)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic Rhinosinusitis With Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | Dupilumab 300 mg (N=143)
Injection Site Erythema (General disorders) | 12 (30) | 8 (25)
Bronchitis (Infections and infestations) | 8 (8) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (25) | 19 (25)
Headache (Nervous system disorders) | 11 (13) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 11 (13)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 17 (26) | 16 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT02912468/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT02912468/SAP_001.pdf